CLINICAL TRIAL: NCT06753019
Title: The Relationship Between The Level of Somatosensory Amplification and Psychological and Functional Status in Patients With Knee Osteoarthritis
Brief Title: Somatosensory Amplification and Psychological and Functional Status In Patients With Knee Osteoarthritis
Status: Recruiting | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mesut ERGAN, Assistant Professor, Suleyman Demirel University
Other Study IDs: 09-27-2024/80/3
Record Dates: First submitted 2024-12-12; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis; Amplification; Kinesiophobia; Psychological Disability; Pain
Keywords: knee osteoarthritis; somatosensory amplification; kinesiophobia; pain; depression
MeSH Terms: conditions — Osteoarthritis, Knee; Kinesiophobia; Pain; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- assessment group: Patients diagnosed with knee OA, who have complaints for at least 6 months, and between the ages of 40-84 will be included in the study.
  Interventions: Other: survey assessment tools

INTERVENTIONS:
Other: survey assessment tools — Functional and psychological status and the level of somatosensory amplification in patients with knee osteoarthritis will be evaluated with questionnaires.

SUMMARY:
As modern society enters the age of an aging population, the prevalence of knee OA continues to increase, which necessitates multi-faceted research. Although there are studies on exaggeration of bodily sensations, depression, kinesiophobia and functional status in patients with knee OA, there are deficiencies in correlating these factors with each other and in directing evaluation and treatment programs. Based on this, this study aims to demonstrate the relationship between the level of exaggeration of bodily sensations, psychological-functional status and perceived pain level in patients with knee pain due to knee OA.

DETAILED DESCRIPTION:
This study is a screening study designed to reveal the relationship between the level of somatosensory amplification and the psychological-functional status and the level of pain felt in patients with knee pain due to knee OA. Considering the correlation of the features to be examined in the literature, it was found that the required sample size should be at least 80 with a test power of 95%, a type I error of 0.05 and an effect size of 0.34. 88 patients between the ages of 40-84 who have been diagnosed with knee OA and have complaints for at least 6 months will be included in the study. Patients with knee pain due to any rheumatologic disease other than OA and individuals with knee pain due to a recent traffic accident or other lower extremity trauma will be excluded from the study. The patients' sociodemographic characteristics such as age, height, weight, body mass index (BMI), gender, education level, marital status will be evaluated using the sociodemographic information form, somatosensory amplification levels will be evaluated with the 'Somatosensory Amplification Scale (SSAS)', the presence of kinesiophobia with the 'Tampa Kinesiophobia Scale (TSK)', pain levels with the Visual Analog Scale (VAS), the presence of depression with the 'Beck Depression Inventory (BDI)', and functional status with the total score of the 'Western Ontario and McMaster Universities Arthritis Index (WOMAC)'. Statistical analysis of the data will be done using IBM SPSS Statistics version 20.0 (SPSS Inc., New York, USA). Kolmogorov-Smirnov test will be used to determine whether the variables are normally distributed, and the socio-demographic information of the participants and the scores they received from the SSAS, TAMPA, VAS, BDI and WOMAC questionnaires will be expressed as percentages, ratios or averages. The linear relationship between quantitative variables will be analyzed with Pearson correlation analysis, and the correlation between qualitative and quantitative variables will be analyzed with variance analysis (ANOVA), and independent samples t-test. In all analyses, p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with knee OA and had complaints for a minimum of 6 months

Exclusion Criteria:

* any rheumatological disease other than OA and individuals with knee pain due to a recent traffic accident or other lower extremity trauma

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suleyman Demirel University Research and Application Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Somatosensory Amplification Scale | up to 2 weeks
  This scale is a 10-item scale developed to measure the magnification/exaggeration that individuals use while somatizing. Each item is scored between 1 and 5. Many of the items include a series of disturbing bodily sensations that are not indicative of illness. The total score is obtained by adding the scores from the items. An increase in the score from the scale indicates that bodily sensations are perceived exaggeratedly.
Tampa Scale for Kinesiophobia | up to 2 weeks
  TSK is a 17-question questionnaire that evaluates fear of re-injury caused by movement, and has been validated and reliable in Turkish. The scale uses a 4-point Likert-type scoring system (1=Strongly disagree, 2=Disagree, 3=Agree, 4=Strongly agree). A total score between 17-68 can be obtained based on the answers given by the person as a result of the questionnaire. A high score indicates a high level of kinesiophobia.
Visual Analog Scale | up to 2 weeks
  The VAS is a 10cm line used to measure the intensity of pain, with 'no pain' at one end and 'extreme pain' at the other. Patients mark the point that best describes their pain intensity. The higher the score, the greater the intensity of pain.
Beck Depression Inventory | up to 2 weeks
  BDI is a scale consisting of 21 questions in total used to determine the level of depression. Each question is evaluated between 0 and 3 points. A total score of 10 and above indicates the presence of depression. 10-18 points indicate minor depression, 19-29 points indicate moderate depression, and 30-63 points indicate severe depression.
Western Ontario and McMaster Universities Arthritis Index | up to 2 weeks
  WOMAC is a 24-item scale developed to evaluate pain, joint stiffness, and physical functions in individuals with knee and hip OA. Total scores range from 0 to 96. A high score on the scale indicates high pain, stiffness, and functional limitations.
sociodemographic data form | up to 2 weeks
  Demographic information (age, height, weight, gender) and socio-cultural (educational status, marital status) data of patients will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: mesut ergan, Study Director — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University Faculty of Health Science, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No